CLINICAL TRIAL: NCT07206628
Title: Real-world Study to Assess Adherence to IOP Lowering Therapy in Glaucoma Patients Using CONNECTDROP®: the GRANITE Study (Glaucoma tReatment AdhereNce wIth connecTed dEvice in Italy)
Brief Title: Real-world Study to Assess Adherence to IOP Lowering Therapy in Glaucoma Patients Using CONNECTDROP®
Status: Recruiting | Type: Observational
Sponsor: Laboratoires Thea (Industry)
Responsible Party: Sponsor
Other Study IDs: LT9060-002
Record Dates: First submitted 2025-09-26; First posted 2025-10-03 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Adherence to Glaucoma Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group receiving T9060 CONNECTDROP

SUMMARY:
The goal of this real-life, national, multicentre, prospective clinical investigation is to describe the adherence rate over time in patients with glaucoma already treated with IOP-lowering eye drops using connected device CONNECTDROP®

The main questions it aims to answer are:

* The mean annual adherence rate, defined as the percentage of the prescribed doses taken by the patient
* The adherence profile of each patient
* The association between the adherence profile, the objective adherence data and the clinical data.

Participants will use the connected device CONNECTDROP® associated with the smartphone application on a daily basis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥ 18 years old), man or woman
* Patient with a diagnosis of bilateral open angle glaucoma
* Patients being prescribed with glaucoma eye drops in EASYGRIP® bottle for at least 6 weeks in monotherapy.
* Patient willing to participate in the study
* Patient who consents for data collection in the frame of the study

Exclusion Criteria:

* Pregnant and/or lactating woman
* Patient receiving another ocular treatment for a chronic condition (i.e. regular instillations for several months)
* Protected patient: adult under guardianship, curatorship or other protection legal, deprived of liberty by judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Glaucoma patients from hospital and/or private practice
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-09-19 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Adherence rate over time in patients with glaucoma already treated with IOP-lowering eye drops in EASYGRIP® bottle clipped with CONNECTDROP® | From enrollment to the end of the study at 12 months
  Assessment of the mean annual adherence rate, defined as the percentage of the prescribed doses actually taken by the patient (i.e. at least 2 instillations per day).

CONTACTS AND LOCATIONS:
Locations (17):
- Italy (17):
  - Besomed SRLS, Bari
  - Studio Oculistico D'Azeglio, Bologna
  - Centro Medico Polispecialistico Di Maita, Catania
  - Studio Medico Oculistico Dr.ssa Rosa SCHIAVELLI s.r.l., Corigliano
  - Ospedale Policlinico S. Martino-IRCCS Clinica Oculistica Università di Genova, Genova
  - Poliambulatorio Chirurgico Modenese Eyecare Clinic, Modena
  - Centro Oculistico Ramovecchi S.r.l., Morrovalle
  - AOU Federico II di Napoli Dipartimento di Neuroscienze e Scienze Riproduttive ed Odontostomatologiche Università degli studi di Napoli Federico II U.O.C. di Oftalmologia, Napoli
  - Azienda Ospedale-Università Padova Ospedale Sant'Antonio UOC Oculistica, Padua
  - A.O.U. Pisana UO Oculistica Universitaria, Pisa
  - Ambulatorio Oculistica Ospedale San Carlo di Nancy -GVM-, Roma
  - Fondazione PTV Policlinico Tor Vergata Fondazione PTV Policlinico Tor Vergata UOSD di Oculistica, Roma
  - IRCCS Fondazione G.B. Bietti per lo Studio e la Ricerca in Oftalmologia ONLUS Presidio Ospedaliero Britannico Unità di Ricerca "Glaucoma, Roma
  - AULSS 4 Veneto Orientale Ospedale di San Donà di Piave Dip. Oculistica, San Donà di Piave
  - AOU Sassari Clinica Oculistica, Sassari
  - Studi Oculistici, Seravezza
  - Humanitas Gradenigo U.O. Oculistica, Torino